CLINICAL TRIAL: NCT06424249
Title: Dynamic Balance in Unilateral Transtibial Amputees Following Virtual Reality Versus Conventional Rehabilitation
Acronym: EQUIL-ARC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Local/2023/EP-02
Record Dates: First submitted 2024-05-16; First posted 2024-05-22 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Amputees / Rehabilitation; Virtual Reality; Postural Balance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality group (Experimental)
  Interventions: Other: Virtual Reality
- Control group (Active Comparator)
  Interventions: Other: Standard rehabilitation

INTERVENTIONS:
Other: Virtual Reality — A progressive rehabilitation protocol (different levels according to success scores) consisting of several exercises using virtual and augmented reality with mechanical perturbations (pitching of the treadmill), interaction with the virtual environment, interaction with the virtual environment and augmented reality (projection of obstacles on the treadmill), and modification of the gait pattern with visual and/or audio biofeedback
  Arms: Virtual Reality group
Other: Standard rehabilitation — A treadmill walking protocol with virtual reality to immerse the patient in a 3 x 5-minute walking session, without visual, mechanical or auditory disturbances, and without prompting the patient to modify their walking pattern.
  Arms: Control group

SUMMARY:
Amputation causes somatic and psychological damage. Prognostic factors for postoperative gait recovery include the need for proprioceptive re-education for dynamic balance. Improved gait patterns and use of the prosthesis contribute to an overall improvement in the amputee's autonomy. Virtual reality coupled with movement analysis allows personalization of treatment with objective assessment of progress.

The study authors hypothesize that a virtual reality protocol for the dynamic balance of a unilateral transtibial amputee in initial rehabilitation will improve the dynamic balance assessment criteria compared with a conventional rehabilitation protocol.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transtibial amputees in hospitalized in the rehabilitation of the musculoskeletal system service
* All etiologies: vascular, traumatic and septic.
* Adapted vascular equipment validated by physician.
* Able to walk for 5 minutes on a treadmill without technical assistance.
* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan

Exclusion Criteria:

* The subject is participating in an interventional study or one involving a drug or medical device, or is in a period of exclusion determined by a previous study
* Patient already included in the present study.
* The subject refuses to or is unable to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Patients with uncorrected or untreated visual disorders.
* Patients with major cognitive disorders (MOCA>23).
* Patients with vestibular disorders.
* Patient with uncontrolled epilepsy.
* Patient with an unhealed amputation stump.
* Patients weighing > 135kg or < 20kg.
* Patients with a functional ambulation category of 1 (i.e. patients requiring the firm, continuous assistance of another person to carry their weight and maintain their balance) or less.
* Patients with medication affecting exercise tolerance,
* Patients with sensory impairments
* Patients with significantly reduced bone density
* Patients for whom it is impossible to correctly adjust the harness to the corresponding body part due to:

  * Body shape
  * Colostomy bags
  * Skin lesions that cannot be adequately protected.
  * Any other reason that prevents proper, pain-free adjustment of the sling.
* Pregnant, parturient or breast-feeding patients.
* Appearance of a stump wound during the study requiring discharge.
* Patient with more than 50% absenteeism from rehabilitation sessions.
* Patient requiring a new prosthesis insert.
* Patient with a serious adverse event affecting dynamic balance rehabilitation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Mediolateral instability during mediolateral external perturbation between groups | Before rehabilitation (Day 1)
  The number of gait cycles required to regain center of mass displacement (number of cycles * cycle time), measured with the GRAIL rehabilitation and movement analysis platform
Mediolateral instability during mediolateral external perturbation between groups | End of rehabilitation sessions (Day 45)
  The number of gait cycles required to regain center of mass displacement (number of cycles * cycle time), measured with the GRAIL rehabilitation and movement analysis platform

SECONDARY OUTCOMES:
Step length variability between groups | Before rehabilitation (Day 1)
  Meters, measured with the GRAIL rehabilitation and movement analysis platform
Step length variability between groups | End of rehabilitation sessions (Day 45)
  Meters, measured with the GRAIL rehabilitation and movement analysis platform
Step width variability between groups | Before rehabilitation (Day 1)
  Meters, measured with the GRAIL rehabilitation and movement analysis platform
Step width variability between groups | End of rehabilitation sessions (Day 45)
  Meters, measured with the GRAIL rehabilitation and movement analysis platform
Cadence variability between groups | Before rehabilitation (Day 1)
  Steps/minute, measured with the GRAIL rehabilitation and movement analysis platform
Cadence variability between groups | End of rehabilitation sessions (Day 45)
  Steps/minute, measured with the GRAIL rehabilitation and movement analysis platform
Center of mass variability between groups | Before rehabilitation (Day 1)
  Meters, measured with the GRAIL rehabilitation and movement analysis platform
Center of mass variability between groups | End of rehabilitation sessions (Day 45)
  Meters, measured with the GRAIL rehabilitation and movement analysis platform
Mobility and balance between groups | Before rehabilitation (Day 1)
  Time Up and Go test, seconds
Mobility and balance between groups | End of rehabilitation sessions (Day 45)
  Time Up and Go test, seconds
Aerobic endurance and functional capacity between groups | Before rehabilitation (Day 1)
  2-minute walk test, meters
Aerobic endurance and functional capacity between groups | End of rehabilitation sessions (Day 45)
  2-minute walk test, meters
Fall risk between groups | Before rehabilitation (Day 1)
  Berg scale, score between 0 and 56 (no fall risk)
Fall risk between groups | End of rehabilitation sessions (Day 45)
  Berg scale, score between 0 and 56 (no fall risk)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Pantera, Principal Investigator — CHU de Nimes
Locations (2):
- France (2):
  - CHU de Nîmes, Hôpital du Grau du Roi, Le Grau-du-Roi
  - CHU de Nimes, Nîmes

IPD SHARING:
Plan to Share IPD: No